CLINICAL TRIAL: NCT05254210
Title: Feasibility Study To Collect Safety And Preliminary Efficacy Data For A Radiofrequency Microneedling Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN20-RF-MN-PROFILES
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Wrinkles; Fine Lines; Crepey Skin; Acne Scars; Active Acne; Enlarged Pores; Loose Skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment with RF Device (Experimental): Subjects may receive up to 3 treatments with the RF device if they are willing to receive treatment for brow lifting and/or present with conditions such as, but not limited to; wrinkles, fine lines, crepey skin, acne scars, active acne, enlarged pores, loose skin on the face, neck and/or body
  Interventions: Device: RF Device (Potenza™)

INTERVENTIONS:
Device: RF Device (Potenza™) — Test spots may be performed prior to the first treatment. Following test spots, for the treatment, the tip will be placed in contact with the skin. Parameters may be adjusted throughout the treatment and will determined by the Clinician.

SUMMARY:
The intended use of the Potenza™ device is to collect clinical data for brow lifting and/or treatment of dermatologic conditions in which electrocoagulation and hemostasis is a viable mechanism for means of improvement.

ELIGIBILITY:
Inclusion Criteria:

* A healthy, non-smoking male or female between the age of 18-60 years old.
* Fitzpatrick skin type I to VI.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 3 months prior to entering this study.
* The subject has a pacemaker.
* The subject had previous use of gold thread skin rejuvenation.
* The subject has a cut, wound, or infected skin on the area to be treated (but skin eruptions may be treated).
* The subject has a metal implant that interferes with the transmission of energy to the electrical field.
* The subject has any embedded electronic devices that give or receive a signal.
* The subject has Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant.
* The subject is allergic to adhesives such as glues on medical tape: they should be alerted that a rash may occur on the neutral electronic monitoring pad (NEM or neutral pad) site, and an over-the-counter preparation may be used to treat the area.
* The subject is allergic to gold.
* The subject has an unrealistic expectation of the results: this is not plastic surgery, and all subjects should be fully informed of the treatment's expected results.
* The subject has nerve insensitivity to heat in the treatment area or in the neutral pad placement area.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated: this treatment will be ineffective.
* The subject has used Accutane (isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it brittle.
* The subject is taking aspirin or are currently taking antiplatelets, thrombolytics, anti-inflammatories or anticoagulants.
* The subject has a history of bleeding coagulopathies.
* The subject is allergic to topical anesthetic.
* The subject has any of the following conditions:

  * Diabetes
  * Epilepsy
  * Autoimmune disease
  * Herpes simplex
  * HIV
  * Hypertension
  * Dermatitis
* The subject has keloid formation propensity.
* Subjects with electronic implants such as cardiac defibrillator. It may interfere with operation of electronic implants or damage the implants, causing risks.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Cautionary Criteria:

* The subject is prone to fever blisters: they should receive a prophylactic antiviral medication regimen prior to treatment.
* The subject has lesions in the treatment area that have not been evaluated and diagnosed: they should be evaluated prior to the treatment day.
* The subject has malignant disease (excluding skin malignancies).
* The subject has used retinoids in the last seven days in the area to be treated: retinoids can create erythema and cause the skin to become heat sensitive.
* The subject has used any chemical peels in the last two to three months in the treatment area: subjects should wait until any remaining erythema or side effects have resolved.
* The subject has tattoos, permanent makeup, and permanent brows in the treatment area: caution must be used. (The ink used in these applications is unregulated and may have metallic components.)
* The subject has a neuropathic disorder, impaired skin sensation or diabetic neuropathy.
* The subject has received fillers or neurotoxin injections: subjects should wait two weeks before receiving a Potenza treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Director of Clinical Research
Locations (1):
- Profiles Beverly Hills, West Hollywood, California, United States

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With RF Device
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With RF Device
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/Persian | 1
  Caucasian | 5
  Brazilian/White | 1
  African American | 2
  Hispanic | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Measure Description: Fitzpatrick Skin Types range from I-VI, with I representing the lowest amount of melanin (lightest skin) and VI representing the highest amount of melanin (darkest skin). Details on this scale can be found in the references section.
  Participants
    Fitzpatrick Skin Type I | 6
    Fitzpatrick Skin Type II | 2
    Fitzpatrick Skin Type III | 0
    Fitzpatrick Skin Type IV | 1
    Fitzpatrick Skin Type V | 1
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Baseline Photographs Compared to Post Treatment Images
Description: Photographs will be evaluated at the baseline and the 30 day follow up. The number of photographs with improvement (based on changes in the skin) from baseline to follow up images will be reported.
Time Frame: 30 day follow up
Population: Each subject had their after picture graded to determine if there was an improvement from the baseline.
Measure: Number; unit: photographs graded as improved
Units Other Than Participants: photographs
Arm/Group | Treatment With RF Device
Number analyzed (Participants) | 8
Number analyzed (photographs) | 8
photographs graded as improved | 8

ADVERSE EVENTS:
Time Frame: Adverse events were captured throughout subject participation in the study, approximately 8 months.
Arm/Group | Treatment With RF Device
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT05254210/Prot_SAP_000.pdf